CLINICAL TRIAL: NCT00956306
Title: A Pharmacokinetic Study of Udenafil in Adult Subjects With or Without Impaired Hepatic Function
Acronym: udenafil
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Dong-A ST Co., Ltd. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DA8159_HI_I
Record Dates: First submitted 2009-08-10; First posted 2009-08-11 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Hepatic Impairment
Keywords: Udenafil,DA-8159,hepatic impairment,healthy volunteers
MeSH Terms: interventions — udenafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Child-Pugh A (Experimental)
  Interventions: Drug: Udenafil
- Child-Pugh B (Experimental)
  Interventions: Drug: Udenafil
- Healthy Volunteers (Experimental)
  Interventions: Drug: Udenafil

INTERVENTIONS:
Drug: Udenafil — 100mg Single Oral Dose of Udenafil
  Other Names: DA-8159; Zydena

SUMMARY:
This study is designed to assess the effect of hepatic impairment on the pharmacokinetics, safety and tolerability of udenafil in subjects with hepatic impairment compared to healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males aged 20 to 64 years at screening.
2. Non-smokers
3. In case of hepatic impaired patients
4. In case of healthy volunteers, the subjects aged ± 10 years old of hepatic impaired patients
5. Subjects within ±20% of the ideal body weight
6. Subjects who have received and understood completely the information regarding the current study and given written informed consents to voluntarily participate in the study and followed all instructions specified in the protocol.

Exclusion Criteria:

1.History of portosystemic shunt surgery.

Ages: 20 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2007-11; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (AUC and Cmax), Safety | up to 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: HYO-SUK LEE, Ph D., Study Chair — Seoul National University Hospital; Young-Suk Lim, Ph D., Principal Investigator — Asan Medical Center, University of Ulsan Colledge of Medicine; Hwi Young Kim, Ph D., Principal Investigator — SMG-SNU Boramae Medical Center; Sook-Hyang Jeong, Ph D., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea